CLINICAL TRIAL: NCT05147246
Title: Catalyzing Change in Education Through a Transformative Learning Collaborative: Scaling-Up of a Social Emotional Learning Curriculum in Uganda
Brief Title: Scaling-Up of a Social Emotional Learning Curriculum in Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-00816
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Social Emotional Learning; Social Emotional Competence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Schools - School Staff (Experimental)
  Interventions: Behavioral: ParentCorps-Professional Development (PD)
- Intervention Schools - Parent-Child Pairs (Experimental)
  Interventions: Behavioral: ParentCorps-Professional Development (PD)
- Wait-List Control Schools - School Staff (No Intervention)
- Wait-List Control Schools - Parent-Child Pairs (No Intervention)

INTERVENTIONS:
Behavioral: ParentCorps-Professional Development (PD) — PD is a school-based evidence-based-intervention (EBI) and preventive service provision model that supports teachers and school personnel to apply EBI strategies to promot young children's medical health in impoverished areas. Teachers and PTAs will participate in a 4-day training before the 1st school term. Teachers in the intervention condition will also receive 8 sessions (8 hours) of face-to-face group-based coaching during the 1st and 2nd terms. Coaching sessions are to help teachers apply EBI strategies in their classrooms, engage families, and develop competencies.
  Arms: Intervention Schools - Parent-Child Pairs; Intervention Schools - School Staff

SUMMARY:
Teachers' social emotional learning/competence (SEL/SEC) can influence teachers' ability in developing healthy teacher-student relationship, managing classroom, implementing evidence-based SEL promotion strategies in classroom, and supporting students' parents. Also, most SEL/SEC interventions have not considered gender equity. Given high prevalence of gender-based violence and high exposure to adverse environment for teachers in low income countries (LIC), which may lead them to greater risk for lower SEC, transforming current education system and considering gender equity and SEL/SEC promotion curriculum to both teachers and children is needed.

The goal of this project is to respond to this need by adapting a locally supported evidence-based-intervention (EBI) for children and further integrates SEL/SEC curriculum for teachers and gender equity component. The EBI to be adapted in this study is ParentCorps-Professional Development (PD), a school-based EBI that trains, empowers, and supports teachers to apply EBI strategies to promote child SEL/SEC and academic learning, and reduce behavioral problems. Two pilot implementation studies from prior work conducted in Uganda and Nepal have demonstrated feasibility, acceptability, usefulness, and efficacy of PD in diverse low resource contexts. PD has shown positive impacts on multiple-level, including positive changes on students' emotional regulation and social competency, teacher-student relationship, and classroom social emotion climate. The proposed research builds on prior positive evidence and further partner with policy and relevant stakeholders to integrate gender equity and teacher SEL/SEC curriculum into the PD (as the PD-Enhance) as well as to test scalable strategies to provide the enhanced PD curriculum at the system level.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the school staff (teachers, head teachers) are: they must be in the recruited study schools and teaching in Pre-Primary to Primary 4 classrooms or holding the head teachers/administration leadership position in school. The inclusion criteria for Parent Leaders are: they must be at least 18 years old and have served as a Parent-Teacher-Association member or Parent Leader in the school for at least 1 year.
* The inclusion criteria for the PD program implementers are: they must have current employment with eligible partners (i.e., medical/mental health institutions, Teacher Training Colleges), with professional experiences in teacher training or mental health training.
* The inclusion criteria for parents are: caregivers must be at least 18 years old, their children must be enrolled in Pre-Primary or Primary 1 to 4 classes (or between 3 to 10 years old) in the recruited schools, and willing to have their child to be assessed by research staff. Parents and children will have diverse characteristics (e.g., randomly selected from school student lists). About 5% families will be randomly selected from the student lists. The proposed study will be open to both men and women caregivers.

Exclusion Criteria:

• Evidence of psychopathology or cognitive impairment severe enough to preclude giving consent, or completing the survey instruments or the focus group of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Number of school staff who displayed a change in teacher EBI practice | 4-6 months post-intervention
Change in Score on Social Competence Scale - Parent (SCP) | Baseline, Month 4-6
  SCP is a 12-item measure that assesses a child's prosocial behaviors, communication skills, and self control. Each item states a behavior that a child may display in a social setting. The parent assesses how well each statement describes the child. Responses are coded on a 5-pt Likert scale: 0=not at all, 1=a little, 2=moderately well, 3=well, and 4=very well. The total score range is 0-48; the higher the score, the better the child is able to regulate his/her emotions.
Change in Score on Difficulties in Emotion Regulation Scale (DERS) - Teacher | Baseline, Month 4-6
  DERS measures emotion dysregulation in an individual. The 18 items, 5 point scale (1=Almost Never, 2=Sometimes, 3=About Half the Time, 4=Most of the Time, 5=Almost Always) yield scores on (a) awareness and understanding of emotions; (b) acceptance of emotions; (c) the ability to control impulses and behave in accordance with goals in the presence of negative affect; and (d) access to emotion regulation strategies that are perceived to be effective for feeling better. The total score range is 18-90; higher scores suggest greater problems with emotion regulation.

SECONDARY OUTCOMES:
Change in Score on Perceived Stress Scale (PSS) - Teacher | Baseline, Month 4-6
  PSS is a 10-question scale that ask about one's feelings and thoughts during the last month. In each case, the teacher is asked to indicate by circling how often he/she felt or thought a certain way. Each question is reported on a 0 (never) - 4 (very often) scale. The total score range is 0-40; the higher the score, the more frequent one has felt stressed.
Change in Score on Patient-Reported Outcomes Measurement Information System (PROMIS) - Anger - Short Form - Parent | Baseline, Month 4-6
  This 5-item form assesses the pure domain of anger in child as reported by parents. The measure is completed by the parent to rate the severity of the child's anger during the past 7 days. Each item is rated on a 5-point scale (1=never to 5=always) with a total score range of 5-25 with higher scores indicating greater severity of anger.
Change in PROMIS - Anxiety - Short Form - Parents | Baseline, Month 4-6
  This 8-item form assesses anxiety in child as reported by parents. The measure is completed by the parent to rate the severity of the child's anxiety during the past 7 days. Each item is rated on a 5-point scale (1=never to 5=always) with a total score range of 8-40 with higher scores indicating greater severity of anxiety.
Change in PROMIS - Depression - Short Form - Parents | Baseline, Month 4-6
  This 6-item form assesses depression in child as reported by parents. The measure is completed by the parent to rate the severity of the i child's depression during the past 7 days. Each item is rated on a 5-point scale (1=never to 5=always) with a total score range of 6-30 with higher scores indicating greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Yen Huang, PhD, MPH, Principal Investigator — NYU Langone Health
Locations (1):
- NAKASEKE, Nakaseke, Uganda

IPD SHARING:
Plan to Share IPD: No
This is a pilot trial of a scale-up model for evidence-based intervention implementation. Given a pilot nature, we are not planning to share the data as public available data. Interested researchers can contact research team for use of the data.